CLINICAL TRIAL: NCT02751398
Title: Impact of Dapagliflozin on DIAstolic Dysfunction in Type 2 Diabetic Patients: The IDDIA Study
Brief Title: Impact of Dapagliflozin on DIAstolic Dysfunction in Type 2 Diabetic Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 4-2015-1130
Record Dates: First submitted 2016-04-14; First posted 2016-04-26 (Estimated); Last update posted 2020-08-11 (Actual); Status verified 2020-08

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — dapagliflozin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dapagliflozin (Experimental): Dapagliflozin 10mg/day
  Interventions: Drug: Dapagliflozin 10mg
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo 10mg

INTERVENTIONS:
Drug: Dapagliflozin 10mg
  Arms: Dapagliflozin
Drug: Placebo 10mg — Matching placebo for dapagliflozin 10 mg
  Arms: Placebo

SUMMARY:
This study aims to assess the impact of 24-week treatment of dapagliflozin in type 2 DM(diabetes mellitus) patients on diastolic dysfunction. Primary endpoint is assessing the impact of 24-week treatment of dapagliflozin in type 2 DM patients on subclinical diastolic dysfunction assessed by supine bicycle diastolic stress echocardiography. Secondary endpoint is assessing the impact of 24-week treatment of dapagliflozin in type 2 DM patients on functional capacity, he impact of 24-week treatment of dapagliflozin in type 2 DM patients at resting diastolic function. This is single-center, randomized, double-blind, placebo-controlled, parallel-arm intervention study.

This study is planned to evaluate the impact of dapagliflozin on diastolic dysfunction assessed. The dose of dapagliflozin will be 10 mg as approved.

For assessment of diastolic dysfunction, supine bicycle stress exercise echocardiography was performed, and changes in diastolic functional reserve, VO2max, exercise time, and maximal exercise capacity were assessed before and after treatment. This study will be randomized, double blind, placebo controlled, to minimize the risk of bias.

ELIGIBILITY:
Inclusion Criteria:

* Female and male aged 19~75 years
* Type 2 DM and had not reached adequate glycemic control with a stable dose of metformin, sulfonylurea, or both drugs before screening
* HbA1c 7.0% ~ 10% at screening (Patients who take metformin only: HbA1C 6.5-10%)
* Patients with ≥ grade 1 diastolic function (relaxation abnormality) at resting echocardiography
* Patients provided with the written, informed consent to participate in this study

Exclusion Criteria:

* Type 1 DM (Fasting c-peptide ≤ 0.78ng/dL(or 0.26 nM/L)), secondary diabetes, gestational diabetes
* History of diabetic ketoacidosis, hyperglycemic hyperosmolar status
* Estimated glomerular filtration rate < 60 mL/min/1.73m2
* History of chronic cystitis or recurrent urinary tract infection
* Currently on loop diuretics
* Currently on medication known to affect glucose metabolism (e.g. corticosteroids, immunosuppressants)
* Abnormal liver function (AST/ALT > x3 upper normal limit)
* On weight loss program or taking weight loss medication
* LV ejection fraction < 50% at resting echocardiography
* Uncontrolled hypertension (systolic blood pressure >200mmHg and/or diastolic blood pressure >110mmHg)
* History of acute myocardial infarction, unstable angina, coronary artery bypass graft or stroke within 6 months
* Inducible ECG abnormalities at exercise
* Cardiomyopathy, significant valvular heart disease, or a significant arrhythmia
* Patients who cannot perform supine bicycle stress echocardiography
* Pregnant or lactating women
* Subjects who the investigator deems inappropriate to participate in this study

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-08-18 (Actual); Primary Completion 2020-06-15 (Actual); Study Completion 2020-06-15 (Actual)

PRIMARY OUTCOMES:
subclinical diastolic dysfunction assessed by supine bicycle diastolic stress echocardiography | 24-week

SECONDARY OUTCOMES:
the impact of dapagliflozin on patients' functional capacity | 24-week
  functional capacity measured by maximum oxygen uptake (VO2max), Exercise time, Maximum exercise capacity (METs)
the impact of dapagliflozin on resting diastolic function | 24-week
  Diastolic function measured by LV mass index, Grade of diastolic function, Ea velocity, Left atrial volume index

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Cardiology, Yonsei Cardiovascular Hospital, Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No